CLINICAL TRIAL: NCT00397605
Title: Cannabinoids in Bipolar Affective Disorder: A Controlled Pilot Study
Brief Title: Cannabinoids in Bipolar Affective Disorder
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: study was never started and no patients were ever enrolled
Sponsor: University of British Columbia (Other)
Collaborators: Vancouver General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: H06-00239
Record Dates: First submitted 2006-11-07; First posted 2006-11-09 (Estimated); Last update posted 2014-09-18 (Estimated); Status verified 2014-09

CONDITIONS: Bipolar Affective Disorder
Keywords: bipolar; therapeutic potential; neurocognitive performance; cannabinoids
MeSH Terms: conditions — Bipolar Disorder

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (1):
- Crossover (Experimental)
  Interventions: Drug: Synthetic cannabinoids (1:1 ratio of THC % CBD)

INTERVENTIONS:
Drug: Synthetic cannabinoids (1:1 ratio of THC % CBD) — Randomized crossover study of 2 weeks of active study medication (maximum daily dosage of 60 mg) vs. 2 weeks of matching placebo.

SUMMARY:
Some people with bipolar disorder who use cannabis (marijuana) claim that it eases the symptoms of depression and mania. There are many chemicals (called cannabinoids) found in cannabis but two particular ones appear to have medicinal (therapeutic) effects. These two compounds are: delta-9-tetrahydrocannabinol (THC) and cannabidiol (CBD). These cannabinoids appear to have mood, anxiety, and sedative effects as well as have antipsychotic and anticonvulsant properties. This study will try to find out if these cannabinoids can be of benefit as an add-on treatment in bipolar disorder and what effects it has on thinking power and memory.

DETAILED DESCRIPTION:
This study will be a within-subject, random order, double-blind cross-over study with standard clinical and neuropsychological ratings. Duration is 13 weeks per subject. Clinical assessments including mood ratings will be performed weekly. Instructions and practice on the use of the spray will be given under supervision during a 2-week run-in period before baseline. Patients can control the dosage of cannabinoids according to their symptoms by administering up to a maximum of 48 pump-controlled sprays per day. Patients will be asked to abstain from using cannabis (other than the study drug) during the study. Patients will be treated for 4 weeks with either the sublingual THC:CBD spray or placebo spray. This will be followed by a 2-week washout period before another 4 weeks of treatment with whichever study medication was not initially used. Neurocognitive testing will be performed 3 times during the study. A mood diary will be completed daily by each patient at home.

ELIGIBILITY:
Inclusion Criteria:

* Outpatients between the 19-60 years of age with a diagnosis of bipolar disorder.
* Women must not be currently pregnant and must use a reliable method of contraception for the duration of the study.
* Subjects must be on stable medication (4 weeks minimum) for their bipolar illness (symptomatic despite current treatment), must be able to provide written informed consent, must adequately understand written and verbal English.

Exclusion Criteria:

* Those not meeting the inclusion criteria and those not able to give informed consent.
* Women who are currently pregnant or nursing.
* Those at immediate risk of harming self or others;
* those who have a clinically significant medical illness or other significant psychiatric illness;
* currently abusing alcohol or drugs;
* currently being treated with an investigational medication or medication that is contraindicated with cannabinoids;
* have a known allergy to cannabis-based products.

Ages: 19 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2006-11; Primary Completion 2013-12 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
To determine whether a standardized plant extract of cannabis containing a 1:1 ratio of THC & CBD can alleviate bipolar mood symptoms unresponsive to standard treatment. To be measured weekly over 13 weeks. | 13 weeks

SECONDARY OUTCOMES:
To determine the effects on cognition.
To be measured at baseline and at the end of each treatment phase.

CONTACTS AND LOCATIONS:
Overall Officials: Allan H. Young, Ph.D, Principal Investigator — University of British Columbia
Locations (1):
- Department of Psychiatry, University of British Columbia, Vancouver, British Columbia, Canada